CLINICAL TRIAL: NCT04169139
Title: A Prospective, Multicenter, Randomized, Blinded and Controlled Study Comparing REPaiR® and MIST Therapies for Treatment of Moderate to Severe Generalized Periodontitis
Brief Title: Controlled Study Comparing REPaiR® and MIST Therapies for Treatment of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGuire Institute (Industry)
Collaborators: Biolase Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOLASE001-2017
Record Dates: First submitted 2019-09-06; First posted 2019-11-19 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: randomized, blinded, parallel arm trial, non-inferiority comparison of REPaiR therapy (experimental treatment) versus MIST (control therapy)
Who Masked: Outcomes Assessor
Masking Description: Examiners are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MIST - minimally invasive surgical therapy (Active Comparator): Beginning with the "papilla preservation technique" (Takei et al), further improved by Cortellini et al (1995) and combined with minimally invasive approaches (Harrel et al 1995), MIST, using "minimally invasive surgical approaches and micro-surgery instruments," has evolved into a decision tree guideline for treating periodontitis based on periodontal pocket morphology and papilla width/ interdental space (Cortellini P, Tonetti MS (2007) J Clin Periodontol;34(1):87-93).
  Interventions: Device: MIST (minimally invasive surgical therapy)
- REPaiR - laser periodontal therapy (Experimental): The REPaiR regimen is a step-by-step protocol for using the Waterlase Express Er,Cr:YSGG laser for periodontitis. The protocol steps and associated laser delivery is controlled by a computer interface that dictates laser tip, energy and associated air and water mixes. Like MIST, REPaiR uses a set, decision tree approach for periodontal therapy, with prescribed steps and laser settings to quantify and standardize treatment. Potential clinical benefit, as with MIST, are not only effective periodontal therapy with reduced recession compared with traditional surgical approaches, but also reduced patient morbidity (Arnabat-Domínguez et al (2010). Lasers Med Sci;25(3):459-64).
  Interventions: Device: MIST (minimally invasive surgical therapy)

INTERVENTIONS:
Device: MIST (minimally invasive surgical therapy) — REPaiR Periodontal Therapy
  Other Names: REPaiR

SUMMARY:
A comparison of laser (REPaiR) compared with minimally invasive surgical therapy for moderate to severe periodontal disease.

DETAILED DESCRIPTION:
The Trial is a multi-center, randomized, blinded, parallel arm trial of REPaiR therapy (experimental treatment) versus MIST (control therapy) in a maximum of 2 qualifying periodontal study teeth will be treated in each subject. Qualifying teeth will have PPD ≥ 6mm and intrabony vertical ≥ 3 mm, with base of defect ≥ 3 mm coronal to the tooth apex, and defect angle ≥ 25°.

For Subjects already in maintenance therapy and having completed scaling and root planing within the previous 6-months, up to 3 Study Teeth will be selected and SRP conducted on just these teeth, and subjects will be randomized to either Test or Control Therapies (Visit 3). For patients already in maintenance therapy and NOT having completed SRP within the previous 6-months, up to 3 qualifying teeth may be selected, and localized SRP in the study teeth quadrants (Visit 2) can be followed after 4-6 weeks by Visit 3 Therapy on up to 2 Study Teeth. Other subjects not in maintenance therapy and with up to 3 qualifying teeth will be selected at the Screening Visit; then 4-6 weeks following SRP, up to 2 Study Teeth will be selected, and subjects will be randomized to either Test or Control Therapies. Follow-up assessments will be conducted on all subjects by a blinded examiner over a 12-month period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 to 75 years of age, inclusive.
* Subjects must be diagnosed with moderate to severe generalized periodontitis (ADA Classification Case Type III or IV) as determined by the investigator.
* Subjects must have at least one, but up to 2, non-adjacent, qualifying Study Teeth with Pockets (PPD ≥ 6 mm & intrabony vertical ≥ 3 mm, with base of defect ≥ 3 mm coronal to the tooth apex, and defect angle ≥ 25° as defined by radiograph) on non-adjacent teeth.
* Subjects will have read, understood and signed an institutional review board (IRB) approved Informed Consent Form (ICF).
* Subjects who are able and willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Visual inability to identify cementoenamel junction (CEJ) or other landmark for probing measures.
* Presence of an acute periodontal abscess at the time of MIST or REPaiR treatment steps
* Mobility > 1 at the time of MIST or REPaiR treatment steps
* Use of 3rd molars, defects distal to terminal 2nd molars, and teeth treated endodontically as study teeth.
* Subjects with healing disorders (such as: diabetes mellitus confirmed HgA1C of > 7 within 6-months of screening, cancer, HIV, bone metabolic diseases or Type IV heart disease) that could compromise wound healing and/ or preclude periodontal surgery; or who are taking medications that compromise wound healing, such as chronic steroid use - either inhaler or systemic, calcium channel blockers with clinical evidence of secondary hyperplastic tissue reactions, anti-seizure medications, medications for bone metabolic diseases, radiation or other immuno-suppressive therapy.
* Traumatic occlusion of study teeth not addressed by occlusal adjustment or splint therapy during the course of the study prior to conclusion of SRP
* Subjects taking intramuscular or intravenous bisphosphonates.
* Subjects smoking >10 cigarettes per day or an equivalent amount of any other nicotine products, such as smokeless chewing tobacco, nicotine patch, vaporizer, gum, pipe, or cigar smoking.
* Female subjects who are pregnant or lactating, or who intend to become pregnant during the study duration.
* Anticipated use of systemic antibiotics during the trial or within 30 days of SRP
* An existing condition that may warrant use of antibiotics during the trial (e.g., ongoing infection noted at Screening Visit, cystic fibrosis or chronic obstructive pulmonary disorder with history of frequent, recurrent lung infections).

Use within 30 days prior to Day 1, or a condition for which use is anticipated during trial: topical oral, nasal and systemic corticosteroids.

* Anticipated use of the agents known to affect periodontal status during the trial and/or use within 30 days prior to Day 1: immunosuppressants, calcium antagonists or phenytoin- - Participation in another clinical study within 90 days prior to Day 1.
* Subjects who received oral health treatments/interventions within 90 days of Day 1, which the investigator believes may interfere with the periodontal parameters to be assessed in this study (e.g., significant dental and/or gum/oral tissue work).
* Untreated moderate to severe periodontitis.
* Subjects, who in the opinion of the Investigator, for any reason other than those listed above, will not be able to complete the study per protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
CAL (Clinical Attachment Level) | 6-months post Sx
  Clinical Attachment Level Measured by Periodontal Probe using PPD and Recession

SECONDARY OUTCOMES:
Radiographic evidence of bone fill | 6-months post Sx
  Standardized periapical radiographs

OTHER OUTCOMES:
Patient Reported Outcome for Pain | Daily for 7-days following Sx
  Patient Reported Outcomes (PROs) for Pain Using 10-Point scale 0-"no pain at all" to 10-"pain as bad as you can imagine" VAS. A low score would indicate a low level of patient reported post-operative pain.
Patient Reported Outcome for Satisfaction | 1-month, 3-months and 6-months post SX
  Satisfaction with Esthetics and Overall Satisfaction with Procedure Using the following list of response options:
  Very satisfied (Scored as 1), Somewhat satisfied (Scored as 2), Neither satisfied nor dissatisfied (Scored as 3), Somewhat dissatisfied (Scored as 4), Very dissatisfied (Scored as 5)
  A low score would indicate a high level of satisfaction with the treatment provided.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Clem, DDS, Principal Investigator — Regenerative Solutions
Locations (1):
- Medelis Inc, Nashville, Tennessee, United States